CLINICAL TRIAL: NCT03801343
Title: Efficacy and Tolerance Evaluation of "Nutrakos®" Amino Acid Food Supplement (Pilot Study)
Brief Title: Efficacy and Tolerance Evaluation of an Amino Acid Food Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1618
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Skin Photoaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrakos® (Experimental): 12 female subjects aged 35-70, have taken during a meal, for the 1 month ,2 stick packs/die of the food supplement
  Interventions: Dietary Supplement: Nutrakos®

INTERVENTIONS:
Dietary Supplement: Nutrakos® — "Nutrakos®" Amino Acid Food Supplement supplies a specific mixture of amino acids that has been proven to induce synthesis of collagen and elastin, the main proteins of derma structure in fibroblasts and keratocytes.

SUMMARY:
Skin moisturizing and elasticizing efficacy of an amino acid food supplement

DETAILED DESCRIPTION:
Primary end point of this study was to evaluate the moisturizing and elasticizing activity of "Nutrakos®" Amino Acid Food Supplement, both photoexposed and not photoexposed on skin areas (forearm volar and dorsal surface) by non-invasive instrumental measurements; the product will be tested for 1 month by female subjects, aged 35-70 years with skin photoaging. An additional aim of this study was to evaluate the product tolerance both by investigator and volunteers.

ELIGIBILITY:
Inclusion Criteria:

* female sex,
* 35-70 years,
* skin phototype II and III according to Fitzpatrick's classification (see par. 8.2.1)
* accepting to not change their habits regarding food, physical activity, body cosmetic and cleansing products;
* accepting not to expose their body to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study;
* accepting to sign the informed consent form.

Exclusion Criteria:

* Pregnancy;
* lactation;
* smokers;
* alcohol or drug abusers;
* skin phototype I, IV, V and VI according to Fitzpatrick's classification
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* subjects not in menopause who do not accept to perform the pregnancy test at T0 and at the end of the study (T1M);
* Body Mass Index (BMI) variation (± 1) during the study period;
* change in the normal habits regarding food, physical activity, body cosmetic and cleansing use during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study currently or during the previous 6 months;
* dermatitis;
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, severe rosacea, scleroderma, local infections and severe acne);
* diabetes;
* endocrine disease;
* hepatic disorder;
* renal disorder;
* cardiac disorder;
* pulmonary disease;
* cancer;
* neurological or psychological disease;
* inflammatory/immunosuppressive disease;
* drug allergy;
* anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year before the study);
* using of drugs able to influence the test results in the investigator opinion.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline of superficial skin hydration | Basal visit (T0), 2 weeks (T2W), 1 month (T1M)
  Skin electrical capacitance value was measured mono-laterally on the right or left forearm (volar and dorsal surface) with Corneometer CM825 (Courage - Khazaka, Köln, Germany). The measure of the skin capacitance properties is an indirect expression of its hydration level.
Change from baseline of deep skin hydration | Basal visit (T0), 2 weeks (T2W), 1 month (T1M)
  Tissue dielectric constant value of superficial and deep skin layers was measured mono-laterally on the right or left forearm (volar and dorsal surface) with MoistureMeterD (Delfin Technologies, Kuopio - Finland)
Change from baseline of skin plastoelasticity | Basal visit (T0), 2 weeks (T2W), 1 month (T1M)
  Superficial and deep skin plastoelasticity were measured mono-laterally on the right or left forearm (volar and dorsal surface) with the instrument Dermal Torque Meter (Dia-Stron Ltd., UK).

SECONDARY OUTCOMES:
Change from baseline of tolerance | Basal visit (T0), 2 weeks (T2W), 1 month (T1M)
  The food supplement tolerance was evaluated considering: any adverse event related to the study treatment, which occurred during the study; any judgement reported by the volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy